CLINICAL TRIAL: NCT02652910
Title: A Two-Arm, Single-Center, Open-Label Pilot Study of IL-2 Programmed or IL-7/IL-15 Programmed Anti-CD19:TCRz:CD28 T-cells in Patient With CD19-Positive Lymphoma That is Resistant or Refractory to Chemotherapy
Brief Title: Memory-enriched CAR-T Cells Immunotherapy for B Cell Lymphoma
Acronym: MeCAR
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Xuzhou Medical University (Other); Hrain Biotechnology Co., Ltd. (Industry); Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Director of Department of Cancer, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20151117
Record Dates: First submitted 2015-11-18; First posted 2016-01-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2016-04

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Follicular Lymphoma; Stage IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IL-2 programmed CD19.CAR-T cells (Experimental): Administrated with IL-2 programmed CD19.CAR-T cells on day 0,1,2 in the lympho-depleted patients
  Interventions: Drug: CD19.CAR-T cells
- IL-7/IL-15 programmed CD19.CAR-T cells (Experimental): Administrated with IL-7/IL-15 programmed CD19.CAR-T cells on day 0,1,2 in the lympho-depleted patients
  Interventions: Drug: CD19.CAR-T cells

INTERVENTIONS:
Drug: CD19.CAR-T cells — Retroviral vector-transduced autologous T cells to express CD19-specific CARs
  Other Names: DSCAR01

SUMMARY:
The goal of this clinical trial is to study how approaches for manufacturing chimeric antigen receptor (CAR)-modified T (CAR-T) cells affect their in vivo persistence and therapeutic efficacy against B lymphoma. Recently, cancer immunotherapy, treatments aiming to arm patients with immunity specifically against cancer cells, has emerged as a promising therapeutic strategy. Among the many emerging immunotherapeutic approaches, clinical trials utilizing CARs against B cell malignancies have demonstrated remarkable potential. CARs combine the variable region of an antibody with T-cell signaling moieties to confer T-cell activation with the targeting specificity of an antibody. Thus, CARs are not MHC-restricted so they are not vulnerable to MHC down regulation by tumors. However, defined by the activation and contraction program of their mother cells, the persistency and function of CAR-T cells are also restricted by the protocol of manufacturing. Previous clinical studies largely utilized interleukin-2 (IL-2) for the ex vivo expansion of CAR-T cells, which preferentially generate CAR-T cells with characteristics of terminally differentiated effector cells. Our preliminary data indicated that two common gamma chain cytokines, IL-7 and IL-15, can help to selectively expand CAR-T cells with various memory phenotypes. CAR-T Cells prepared under this condition resulted in improved therapeutic efficacy in preclinical animal models. This clinical investigation is to test a hypothesis whether IL-7/IL-15-programmed anti-CD19 CAR-T cells persist longer in lymphoma patients after infusion and whether the persistency of CAR-T cells can lead to improved anti-lymphoma efficacy.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the safety and feasibility of CD19.CAR-T cells manufactured through IL-7/IL-15-mediated expansion or IL-2-mediated expansion
2. To determine in vivo dynamics and persistency of IL-7/IL-15 programmed CD19.CAR-T cells.
3. To determine the efficacy of IL-7/IL-15 programmed CD19.CAR-T cells in treating patients with CD19-positive lymphoma

Secondary Objectives

1. To determine whether the IL-7/IL-15 programmed CD19.CAR-T cells are superior to the IL-2 programmed cells as measured by their in vivo persistence post infusion
2. To determine whether the IL-7/IL-15 programmed CD19.CAR-T cells are superior to the IL-2 programmed cells as measured by their efficacy in lymphoma therapy
3. To assess the dynamics of intratumoral infiltration of CD19.CAR-T cells.
4. To correlate the subsets and differentiation of CD19.CAR-T cells to observed anti-tumor efficacy

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years to 70 Years, Male and female;
2. Expected survival > 12 weeks;
3. Performance score 0-2;
4. Histologically confirmed as CD19-positive lymphoma and who meet one of the following conditions;

   * Patient receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment;
   * Disease recurrence after stem cell transplantation;
   * Diagnosis as lymphoma, but refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy
5. Creatinine < 2.5 mg/dl;
6. ALT/AST < 3x normal;
7. Bilirubin < 2.0 mg/dl;
8. Adequate venous access for apheresis, and no other contraindications for leukapheresis;
9. Take contraceptive measures before recruit to this trial;
10. Written voluntary informed consent is given.

Exclusion Criteria:

1. Patients with symptoms of central nervous system
2. Accompanied by other malignant tumor
3. Active hepatitis B or C, HIV infection
4. Any other diseases could affect the outcome of this trial
5. Suffering severe cardiovascular or respiratory disease
6. Poorly controlled hypertension
7. A history of mental illness and poorly controlled
8. Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration
9. Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
10. Reaching a steady dose if receiving anticoagulant therapy before assignment
11. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
12. Pregnant or lactating women
13. Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 4 weeks
Phase 2: Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 8 weeks
Phase 2: Comparison of overall complete remission rate for the two arms | One year

SECONDARY OUTCOMES:
Duration of remission | One year
Minimum residual disease negative remission rate | 8 weeks
Duration of CAR-positive T cells in circulation | 6 months
Total number of CAR-positive T cells infiltrated into lymphoma tissue | 6 months
Overall survival | One year

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zhu, M.D., Ph.D., Principal Investigator — Department of Cancer of Xinqiao Hospital
Locations (1):
- Department of Oncology, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338